CLINICAL TRIAL: NCT06262347
Title: NIDA CTN Protocol 0150: Personally-Tailored Opioid-overdose and Medication for Opioid Use Disorder (MOUD) Education (TOME) for Pregnant and Postpartum Persons in MOUD: A Pilot Randomized Trial (TOME Trial)
Brief Title: Personally-Tailored Opioid-overdose and Medication for Opioid Use Disorder (MOUD) Education (TOME) for Pregnant and Postpartum Persons in MOUD
Acronym: TOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: T. John Winhusen, PhD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, T. John Winhusen, PhD, Professor; Vice Chair and Division Director of Addiction Sciences, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0115; UG1DA013732 (NIH)
Record Dates: First submitted 2024-02-05; First posted 2024-02-16 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Opioid Use Disorder; Pregnancy Related; Substance Use; Drug Abuse; Drug Abuse in Pregnancy; Drug Addiction
Keywords: CTN-0150; clinical trials network
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Dosage Forms; Educational Status

STUDY DESIGN:
Intervention Model Description: This is an intent-to-treat, two-arm, open-label, randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personally-Tailored Opioid-overdose and Medication for opioid use disorder (MOUD) Education (TOME) (Experimental): Drug: Naloxone kit
  Naloxone nasal spray (NARCAN) is a potentially life-saving medication that can stop or reverse the effects of an opioid overdose. This nasal spray is approved by the FDA for reversing OODs and has a favorable side-effects profile. A take-home kit will be provided to participants, which may be useful in the event of a future opioid overdose.
  Behavioral: Personally-Tailored Opioid-overdose and Medication for opioid use disorder (MOUD) Education (TOME)
  TOME entails a trained RA: 1) administering a REDCap survey to assess an individual's opioid-overdose/MOUD knowledge; and 2) reviewing the personal feedback reports with the recipient.
  Interventions: Behavioral: Personally-Tailored Opioid-overdose and Medication for opioid use disorder (MOUD) Education (TOME)
- Control (Active Comparator): Drug: Naloxone kit
  Naloxone nasal spray (NARCAN) is a potentially life-saving medication that can stop or reverse the effects of an opioid overdose. This nasal spray is approved by the FDA for reversing OODs and has a favorable side-effects profile. A take-home kit will be provided to participants, which may be useful in the event of a future opioid overdose.
  Behavioral: SAMHSA handouts
  SAMHSA handouts: 1) "Opioid Overdose Prevention Toolkit: Safety Advice for Patients and Family Members"; 2) "Opioid Overdose Prevention Toolkit: Recovering from Opioid Overdose"; and 3) "Medication-Assisted Treatment for Opioid Addiction: Facts for Families and Friends". These handouts can be offered as physical copies or electronically.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Personally-Tailored Opioid-overdose and Medication for opioid use disorder (MOUD) Education (TOME) — The TOME intervention is a modified version of the personally-tailored opioid overdose prevention education and naloxone distribution (PTOEND) intervention (Winhusen et al. Evaluation of a personally-tailored opioid overdose prevention education and naloxone distribution intervention to promote harm reduction and treatment readiness in individuals actively using illicit opioids. Drug Alcohol Depend. Nov 1 2020;216:108265). Modifications include updating the knowledge assessment/education to reflect changes in the drug supply (i.e., the current high prevalence of fentanyl and increasing prevalence of xylazine) and the addition of items specific to pregnancy. Like PTOEND, TOME is a computer-guided intervention which utilizes REDCap to complete assessments and automatically generate personally-tailored feedback reports.
  Arms: Personally-Tailored Opioid-overdose and Medication for opioid use disorder (MOUD) Education (TOME)
Behavioral: Control — Participants randomized to the control condition will be offered three SAMHSA handouts.
  Arms: Control

SUMMARY:
The primary objective of this study is to evaluate the ability of TOME to increase Medication for Opioid Use Disorder (MOUD) and opioid-overdose knowledge in pregnant and postpartum persons.

DETAILED DESCRIPTION:
This is an intent-to-treat, two-arm, open-label, randomized controlled trial. Eligible participants will be randomized in a 1:1 ratio to TOME or Control, balancing on site. Participants will receive the assigned intervention following randomization and will complete a three week follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

Potential participants must be:

1. 18 years of age or older;
2. Pregnant or be within 12 months postpartum;
3. Enrolled in MOUD (either buprenorphine or methadone) at the study site or affiliated clinic where enrollment can be confirmed;
4. Able to understand the study, and having understood, provide written informed consent in English

Exclusion Criteria:

Potential participants must not:

1. have suicidal or homicidal ideation requiring immediate attention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T. John Winhusen, PhD, Principal Investigator — University of Cincinnati
Locations (6):
- United States (6):
  - Gateway Community Services, Jacksonville, Florida
  - Pregnancy Recovery Center at Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah SUPeRAD Clinic, Salt Lake City, Utah
  - Marshall Health MARC Program, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Primary data for this study will be available to the public in the NIDA data repository, per NIDA CTN policy.
Supporting Information: Study Protocol
URL: https://datashare.nida.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Personally-Tailored Opioid-overdose and Medication for Opioid Use Disorder (MOUD) Education (TOME): Drug: Naloxone kit
  TOME: Each participant's knowledge of Medication for Opioid Use Disorder (MOUD) and opioid-related overdose (OOD) was assessed. A trained research assistant met individually with the participant for ≤15 minutes to review incorrect answers and explain the correct answers using four computer-generated feedback reports: 1) MOUD; 2) OOD risk factors; 3) signs of an OOD; and 4) how to respond to an OOD. Participants were offered a copy of their personal feedback reports.
- Control: Drug: Naloxone kit
  Naloxone nasal spray (NARCAN) is a potentially life-saving medication that can stop or reverse the effects of an opioid overdose. This nasal spray is approved by the FDA for reversing OODs and has a favorable side-effects profile. A take-home kit will be provided to participants, which may be useful in the event of a future opioid overdose.
  Behavioral: SAMHSA handouts
  SAMHSA handouts: 1) "Opioid Overdose Prevention Toolkit: Safety Advice for Patients and Family Members"; 2) "Opioid Overdose Prevention Toolkit: Recovering from Opioid Overdose"; and 3) "Medication-Assisted Treatment for Opioid Addiction: Facts for Families and Friends". These handouts can be offered as physical copies or electronically.
  Control: Participants randomized to the control condition will be offered three SAMHSA handouts.
Period: Overall Study
Arm/Group | Personally-Tailored Opioid-overdose and Medication for Opioid Use Disorder (MOUD) Education (TOME) | Control
Started | 67 | 64
Completed | 63 | 60
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Personally-Tailored Opioid-overdose and Medication for Opioid Use Disorder (MOUD) Education (TOME): Drug: Naloxone kit
  Naloxone nasal spray (NARCAN) is a potentially life-saving medication that can stop or reverse the effects of an opioid overdose. This nasal spray is approved by the FDA for reversing OODs and has a favorable side-effects profile. A take-home kit will be provided to participants, which may be useful in the event of a future opioid overdose.
  Behavioral: TOME
  TOME: Each participant's knowledge of Medication for Opioid Use Disorder (MOUD) and opioid-related overdose (OOD) was assessed. A trained research assistant met individually with the participant for ≤15 minutes to review incorrect answers and explain the correct answers using four computer-generated feedback reports: 1) MOUD; 2) OOD risk factors; 3) signs of an OOD; and 4) how to respond to an OOD. Participants were offered a copy of their personal feedback reports.
- Total: Total of all reporting groups
Arm/Group | Personally-Tailored Opioid-overdose and Medication for Opioid Use Disorder (MOUD) Education (TOME) | Control | Total
Number analyzed (Participants) | 67 | 64 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 64 | 131
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (5.0) | 30.7 (4.8) | 31.2 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 64 | 131
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 64 | 57 | 121
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 58 | 59 | 117
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Medication for Opioid Use Disorder (MOUD) Knowledge Score [Mean (Standard Deviation); unit: percentage of correct answers] — This outcome is measured by the Opioid Overdose and Treatment Awareness Survey (OOTAS) knowledge evaluation:
  MOUD knowledge, potential score of 0-10; higher score indicates more knowledge. Values are converted to a percentage of correct answers from 0-100% where higher percentages mean more knowledge.
  percentage of correct answers | 64.0 (15.4) | 69.5 (12.1) | 66.7 (14.1)
Opioid Overdose Knowledge Score [Mean (Standard Deviation); unit: percentage of correct answers] — This outcome is measured by the first three sections of the Opioid Overdose and Treatment Awareness Survey (OOTAS).
  Opioid-overdose knowledge, potential score of 0-31; higher score indicates more knowledge. Values are converted to a percentage of correct answers from 0-100% where higher percentages mean more knowledge.
  percentage of correct answers | 81.7 (7.1) | 82.5 (5.6) | 82.1 (6.4)
Medication for Opioid Use Disorder (MOUD) Internalized Stigma [Mean (Standard Deviation); unit: average score] — This will be assessed with the The Methadone Maintenance Treatment Stigma Mechanisms Scale (MMT-SMS) questionnaire.
  Score range: 1 - 5; higher score indicates greater MOUD stigma
  average score | 1.8 (0.7) | 1.7 (0.8) | 1.7 (0.8)
Drug Self-efficacy [Mean (Standard Deviation); unit: average score] — This will be assessed with the Thoughts about abstinence (TAA) instrument. Drug Self-efficacy Score range: 0 - 9; higher score indicates greater expected success in avoiding drug use
  average score | 2.6 (2.6) | 2.7 (2.9) | 2.6 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Medication for Opioid Use Disorder (MOUD) Knowledge Score
Description: This outcome is measured by the Opioid Overdose and Treatment Awareness Survey (OOTAS) knowledge evaluation:
  MOUD knowledge, potential score of 0-10; higher score indicates more knowledge. Values are converted to a percentage of correct answers from 0-100% where higher percentages mean more knowledge.
Time Frame: Week 3
Population: Several participants were lost to follow-up, explaining why the Week 3 participant numbers analyzed differs from the overall.
Measure: Mean (Standard Deviation); unit: percentage of correct answers
Arm/Group | Personally-Tailored Opioid-overdose and Medication for Opioid Use Disorder (MOUD) Education (TOME) | Control
Number analyzed (Participants) | 63 | 60
percentage of correct answers | 83.5 (15.6) | 72.0 (14.2)

2. Primary Outcome: Opioid Overdose Knowledge Score
Description: This outcome is measured by the first three sections of the Opioid Overdose and Treatment Awareness Survey (OOTAS).
  Opioid-overdose knowledge, potential score of 0-31; higher score indicates more knowledge. Values are converted to a percentage of correct answers from 0-100% where higher percentages mean more knowledge.
Time Frame: Week 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of correct answers
Arm/Group | Personally-Tailored Opioid-overdose and Medication for Opioid Use Disorder (MOUD) Education (TOME) | Control
Number analyzed (Participants) | 63 | 60
percentage of correct answers | 90.1 (7.6) | 82.6 (6.2)

3. Secondary Outcome: Medication for Opioid Use Disorder (MOUD) Internalized Stigma
Description: This will be assessed with the The Methadone Maintenance Treatment Stigma Mechanisms Scale (MMT-SMS) questionnaire.
  Score range: 1 - 5; higher score indicates greater MOUD stigma
Time Frame: Week 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: average score
Arm/Group | Personally-Tailored Opioid-overdose and Medication for Opioid Use Disorder (MOUD) Education (TOME) | Control
Number analyzed (Participants) | 63 | 60
average score | 1.5 (0.7) | 1.6 (0.8)

4. Secondary Outcome: Drug Self-efficacy
Description: This will be assessed with the Thoughts about abstinence (TAA) instrument.
  Drug Self-efficacy Score range: 0 - 9; higher score indicates greater expected success in avoiding drug use
Time Frame: Week 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: average score
Arm/Group | Personally-Tailored Opioid-overdose and Medication for Opioid Use Disorder (MOUD) Education (TOME) | Control
Number analyzed (Participants) | 63 | 60
average score | 2.3 (2.9) | 1.9 (2.6)

ADVERSE EVENTS:
Time Frame: Consent through Week 3
Description: Staff assessed for two AEs that would be of clinical import: 1. Suicidal ideation and 2. Homicidal ideation. SAEs were only reported for events related to a study-defined AE (e.g., hospitalization due to suicidal ideation, etc.).
Arm/Group | Personally-Tailored Opioid-overdose and Medication for Opioid Use Disorder (MOUD) Education (TOME) | Control
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/64
Other Adverse Events (participants affected / at risk) | 0/67 | 0/64

LIMITATIONS AND CAVEATS:
A significant limitation is that the participant sample was primarily White (89.3%) and non-Latino (92.4%) and, thus, it is unknown whether the results would generalize to a more racially and ethnically diverse population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT06262347/Prot_SAP_001.pdf
  • Informed Consent Form (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT06262347/ICF_000.pdf